CLINICAL TRIAL: NCT00373061
Title: The Xolair® Pregnancy Registry: An Observational Study of the Use and Safety of Xolair® (Omalizumab) During Pregnancy
Brief Title: An Observational Study of the Use and Safety of Xolair® During Pregnancy
Acronym: EXPECT
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: Q2952g
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pregnant Women Exposed to Xolair®: Women who are exposed to at least one dose of Xolair® within 8 weeks prior to conception or at any time during their pregnancy will be followed to completion of their pregnancies.
  Interventions: Drug: Xolair®

INTERVENTIONS:
Drug: Xolair® — This being an observational study, the study protocol does not specify any dose regimen.
  Other Names: Omalizumab

SUMMARY:
The Xolair® Pregnancy Registry is an observational study established by Genentech to obtain data on pregnancy outcomes in women who are exposed to Xolair®. Women exposed to at least one dose of Xolair® within 8 weeks prior to conception or at any time during their pregnancy will be followed to completion of their pregnancies. The evaluation of infants will be conducted at birth and at 6-month intervals until the infants are 12 months old. Follow-up of the infant will be extended until the infant is 18 months old, if the woman continues Xolair® treatment while breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

- Women who have been exposed to at least one dose of Xolair® (whether inadvertent or deliberate) within 8 weeks prior to conception or during pregnancy

Exclusion Criteria:

* Women not currently pregnant
* Women exposed to Xolair® not during pregnancy but only while breastfeeding
* Re-enrollment of women who are pregnant for second (or more) time is not allowed

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women exposed to at least one dose of Xolair® within 8 weeks prior to conception or at any time during their pregnancy. Enrollment in the Xolair® Pregnancy Registry is voluntary and must be initiated by the pregnant woman. A healthcare provider cannot enroll a patient but can suggest that the pregnant woman call the Registry Center to enroll herself.
Sampling Method: Non-Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2006-10-20 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Number of Live Births | At Delivery (up to approximately 9 months after enrollment)
Number of Elective Terminations | At Delivery (up to approximately 9 months after enrollment)
Number of Fetal Deaths or Stillbirths | At Delivery (up to approximately 9 months after enrollment)
Number of Congenital Birth Anomalies | At Delivery (up to approximately 9 months after enrollment)

SECONDARY OUTCOMES:
Number of Spontaneous Abortions | At Delivery (up to approximately 9 months after enrollment)
Number of Pregnancy Complications or Abnormalities | Up to approximately 9 months after enrollment
Number of Delivery Complications or Abnormalities | At Delivery (up to approximately 9 months after enrollment)
Gestational Age of Neonates/Infants | Up to approximately 9 months after enrollment
Apgar Score of Neonates/Infants | Delivery (up to approximately 9 months after enrollment) to 18 months
Number of Infant Illnesses or Infections | Delivery (up to approximately 9 months after enrollment) to 18 months
Neonatal Platelet Count | Delivery (up to approximately 9 months after enrollment) to 18 months
Weight of Neonates/Infants | At Delivery (up to approximately 9 months after enrollment)
Length of Neonates/Infants | At Delivery (up to approximately 9 months after enrollment)
Head Circumference of Neonates/Infants | At Delivery (up to approximately 9 months after enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Hoffmann-La Roche, Study Director — Hoffmann-La Roche
Locations (1):
- Ppd Development, Llc, Morrisville, North Carolina, United States